CLINICAL TRIAL: NCT06810687
Title: Is Methenamine Prophylaxis for Urinary Tract Infection After Midurethral Sling as Effective as Antibiotic Prophylaxis? A Randomized Controlled Trial
Brief Title: Is Methenamine Prophylaxis for Urinary Tract Infection After Midurethral Sling as Effective as Antibiotic Prophylaxis?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Shaun Adair, MD, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2248168-1
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infection (Diagnosis)
Keywords: urinary tract infection; midurethral sling; prophylaxis; methenamine
MeSH Terms: conditions — Urinary Tract Infections; Disease | interventions — methenamine hippurate; Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methenamine prophylaxis (Experimental): Methenamine will be prescribed for urinary tract infection prophylaxis
  Interventions: Drug: Methenamine Hippurate 1g BD
- Antibiotic prophylaxis (Active Comparator): Antibiotic prophylaxis chosen per physician preference
  Interventions: Other: Antibiotic prophylaxis

INTERVENTIONS:
Drug: Methenamine Hippurate 1g BD — Antibiotic prophylaxis
  Arms: Methenamine prophylaxis
Other: Antibiotic prophylaxis — Antibiotic prophylaxis
  Arms: Antibiotic prophylaxis

SUMMARY:
Stress urinary incontinence (SUI) affects at least 40% of women in the United States. Synthetic polypropylene mid-urethral slings (MUS) are the gold standard treatment for SUI. Post-operative urinary tract infections (UTI) are one of the most common complications after MUS placement. Some studies have demonstrated that MUS placement can increase the risk of UTI up to 21-34%.

Post-operative UTI can lead to significant healthcare and patient burden. This additional burden further contributes to an estimated annual cost of $1.6 billion for UTI management in the United States. With increased antibiotic usage, there is simultaneous increase in bacterial resistance leading to treatment refractory UTI.

The investigators prescribe post-operative antibiotics prophylactically for 3 days after MUS placement with or without concurrent pelvic reconstructive surgery based on prior literature recommending post-operative prophylaxis. There is a greater emphasis on limiting antibiotic use given the trend of development of bacterial resistance. There are studies supporting alternatives such as methenamine for recurrent UTI prophylaxis treatment, but there are limited studies evaluating methenamine for UTI prophylaxis after MUS.

DETAILED DESCRIPTION:
Synthetic polypropylene mid-urethral slings (MUS) are the gold standard for treatment of stress urinary incontinence (SUI). The most common post-operative complications are urinary tract infection (UTI), bladder injury, bleeding, and mesh erosion. Amongst these complications, post-operative urinary tract infections are the most common complication with incidences up to 21-34%. With high incidences in post-operative UTI, previous studies have shown evidence for the use of prophylactic antibiotics after MUS placement. Previous studies have demonstrated prophylactic antibiotics after MUS placement decreased the incidence of post-operative UTI in the treated groups. While the use of post-operative prophylactic antibiotics may decrease the risk of post-operative UTI, it is essential to consider the broader implication of such antibiotic use.

Along with increased antibiotic use, there is an increase in multidrug resistant uropathogens. This has led to an increased emphasis on antibiotic stewardship to optimize patient care by minimizing the risk of developing antibiotic resistant organisms, preserving effectiveness of currently used antibiotics, and promoting appropriate prescribing practices. There are no studies evaluating post-operative UTI prophylaxis after MUS with methenamine.

Methenamine is a urinary antiseptic that acts when methenamine is converted to ammonia and formaldehyde, which denatures bacterial proteins and nucleic acids. There is no evidence of bacterial resistance to methenamine. Methenamine has been shown to be non-inferior to antibiotic prophylaxis in the setting of recurrent UTI. Methenamine has most commonly been used as long-term UTI prophylaxis treatment, but there are studies demonstrating benefit from short-term methenamine use for prophylaxis.

The investigator's aim is to evaluate whether methenamine is non-inferior to antibiotic prophylaxis after MUS procedure in preventing post-operative UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age ≥ 18
3. Patients undergoing mid-urethral sling procedure

Exclusion Criteria:

1. Medication intolerance or allergy to study medications
2. Renal impairment with GFR <30
3. Breast feeding
4. Pregnancy
5. Recurrent urinary tract infections
6. Active urinary tract infection
7. Immunosuppressive disease
8. Interstitial cystitis

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary tract infection | Within 6 weeks after the procedure
  Urinary tract infection (Positive urine culture) within 6 weeks post-operatively after completing 3 days of antibiotics or methenamine

SECONDARY OUTCOMES:
Number of participants with adverse effects | within 6 weeks after the procedure
  Adverse effects or side effects of treatment
Occurrence of additional treatment of UTI | Within 6 weeks after the procedure
  Further treatment antibiotics given to participants

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No